CLINICAL TRIAL: NCT01899911
Title: Pulse Oximeter Response TO Multiple Levels Of Stable Hypoxia
Brief Title: Clinical Study of Peripheral Capillary Oxygen Saturation (SpO2): Vital Signs Patch (VSP)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: LifeWatch Services, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CD-0024
Record Dates: First submitted 2013-07-07; First posted 2013-07-16 (Estimated); Results first posted 2015-08-28 (Estimated); Last update posted 2015-08-28 (Estimated); Status verified 2015-08

CONDITIONS: Desaturation of Blood

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Vital Signs Patch (VSP) (Experimental): Infrared and Red absorbance measurement on chest
  Interventions: Device: Vital Signs Patch (VSP)

INTERVENTIONS:
Device: Vital Signs Patch (VSP) — Infrared and red absorbance measurement
  Other Names: Vital signs Patch; VSP

SUMMARY:
A clinical study designed to determine the accuracy of the peripheral capillary oxygen saturation (SpO2) function of the Vital Signs Patch (VSP) device for measuring blood saturation level.

DETAILED DESCRIPTION:
The clinical study protocol was designed for determining the accuracy of the SpO2 function of the Vital Signs Patch device for measuring blood oxygen saturation level, according to the guidelines for "evaluating and documenting SpO2 accuracy in human subjects" as set out in Annex EE of ISO 80601-2-61. Section 4.

ELIGIBILITY:
Inclusion Criteria:

* Ages 23 to 33.
* Skin tone varied from light to dark.

Exclusion Criteria:

* Smokers
* Anemic

Ages: 23 Years to 33 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2013-03; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philip E., Bickler, Ph.D., M.D., Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, Room M454, Moffitt Hospital, Box 0542, UCSF,, San Francisco, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Vital Signs Patch (VSP): Infrared and Red absorbance measurement on chest
  VSP: Infrared and red absorbance measurement
Period: Overall Study
Arm/Group | Vital Signs Patch (VSP)
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Vital Signs Patch (VSP)
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Composite Outcome Measure: Successful Capture of Peripheral Capillary Oxygen Saturation (SpO2) Level
Description: Successful capture of SpO2 levels - Infrared and red light absorbency was measured and used for SpO2 percentage calculation from both the Vital Signs Patch (VSP) study device and an invasive Blood Arterial Hemoximeter (standard method) to determine the level of accuracy of data obtained from the VSP device when compared data taken from the Arterial Hemoximeter. A comparison was made by calculating the Average Root Mean Square (Arms) and comparing against the Arms error rate limit of less than or equal to 3.5% at a 95% confidence level. The outcome is either positive or negative - this is a composite outcome measure.
Time Frame: within 24 hrs
Population: Peripheral capillary oxygen saturation (SpO2) Measurements Taken on the 12 Participants
Measure: Number; unit: participants
Arm/Group | Vital Signs Patch (VSP)
Number analyzed (Participants) | 12
participants | 12

ADVERSE EVENTS:
Time Frame: Adverse event collection was limited to the duration of the study for each participant, which was 24 hours.
Description: No adverse event data was observed during the performance of the study.
Arm/Group | Vital Signs Patch (VSP)
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 0/12

LIMITATIONS AND CAVEATS:
Not applicable for this trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less